CLINICAL TRIAL: NCT04970953
Title: Prospective Analysis of Diastolic Stress Tests to Detect Exercise Induced Heart Failure With Preserved Ejection Fraction (HFpEF) in Patients With Intermediate Risk (DEST-HF Study, Diastolic Exercise Stress Testing in Heart Failure)
Brief Title: Diastolic Exercise Stress Testing in Heart Failure
Acronym: DEST-HF
Status: Terminated | Type: Observational
Why Stopped: We raised ethical concerns to proceed an invasive study despite having shown the expected results after 19 patients.
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Peter Lüdike, Professor of Cardiology, University Hospital, Essen
Other Study IDs: 21-9993-BO
Record Dates: First submitted 2021-07-07; First posted 2021-07-21 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: diastolic stress testing; HFpEF

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with intermediate risk for HFpEF at rest: Patients with a HFA-PEFF score of 2-4 points and no obvious extracardiac explanation for exercise-induced dyspnea. Right heart catheterization with be performed at rest and during stress testing.
  Interventions: Procedure: Right heart catheterization

INTERVENTIONS:
Procedure: Right heart catheterization — Right heart catheterization will be performed via a brachial access under sonographic guidance and hemodynamic measurements will be performed in a semi-supine position.

SUMMARY:
Patients with an intermediate risk (HFA-PEFF score 2-4 points) for heart failure with preserved ejection fraction (HFpEF) will be further investigated with invasive right heart catheterization. All patients with a resting pulmonary artery wedge pressure (PAWP) <15mmHg will undergo the following stress test modalities in a randomized order: (1) bicycle ergometry, (2) dynamic handgrip exercise, (3) 500ml fluid challenge over 5 minutes, (4) leg raise testing. Exercise induced HFpEF will be diagnosed if PAWP rises to >25mmHg.

DETAILED DESCRIPTION:
Patients reporting to the investigators' clinic for in- and outpatient consultation and a HFA-PEFF score of 2-4 points will be recruited if their dyspnea is not sufficiently explained by other causes than HFpEF. Patients will undergo a baseline clinical exam, transthoracic echocardiography with measurement of diastolic parameters, and ECG. NYHA class will be reported, standard lab works (NTproBNP, GFR, CRP, Hb, PLT, blood gas analysis) will be taken. The number of patients with a PAWP increase in right heart catheterization (brachial access under sonographic guidance) from a resting value of <15mmHg to >25mmHg during stress testing will be assessed across the four interventions. During bicycle ergometry (semi-supine position) spiroergometric data and gas exchange variables (cardiopulmonary exercise testing) will be co-assessed. Between the testing modalities a 10-minute break will allow hemodynamic variables to normalize.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Unclear etiology of dyspnea with non-invasive testing
* HFA-PEFF score 2-4 points and thus an intermediate risk for HFpEF
* Willingness to participate and obtained written consent

Exclusion Criteria:

* Consent for study participation not obtained
* Age < 18 years
* Medical contraindications to perform right heart catheterization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients reporting to the investigators' in- and outpatient clinic with unsolved dyspnea through non-invasive testing and a HFA-PEFF score 2-4 points and thus an intermediate risk for HFpEF. Following the diagnostic algorithm of HFpEF invasive stress testing is indicated.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
PAWP increase across the four stress tests | 1 year
  Number of patients with an increase of PAWP<15mmHg at rest to >25mmHg during stress testing.

SECONDARY OUTCOMES:
Changes of mean pulmonary artery pressure (mPAP) across the four stress tests | 1 year
  mPAP changes [mmHg] during stress testing will be assessed.
Association of PAWP increase and changes of VO2peak during bicycle ergometry | 1 year
  associations between PAWP [mmHg] and VO2peak [ml/kg/min] during bicycle ergometry will be assessed.
Changes of pulmonary vascular resistance (PVR) across the four stress tests | 1 year
  PVR changes [WU, Wood Units] during stress testing will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lüdike, Professor, Principal Investigator — University Hopsital Duisburg-Essen
Locations (1):
- Klinik für Kardiologie und Angiologie-Westdeutsches Herz- und Gefäßzentrum Essen, Essen, Nordrhein, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pieske B, Tschope C, de Boer RA, Fraser AG, Anker SD, Donal E, Edelmann F, Fu M, Guazzi M, Lam CSP, Lancellotti P, Melenovsky V, Morris DA, Nagel E, Pieske-Kraigher E, Ponikowski P, Solomon SD, Vasan RS, Rutten FH, Voors AA, Ruschitzka F, Paulus WJ, Seferovic P, Filippatos G. How to diagnose heart failure with preserved ejection fraction: the HFA-PEFF diagnostic algorithm: a consensus recommendation from the Heart Failure Association (HFA) of the European Society of Cardiology (ESC). Eur Heart J. 2019 Oct 21;40(40):3297-3317. doi: 10.1093/eurheartj/ehz641. PMID 31504452